CLINICAL TRIAL: NCT06772818
Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics of the Nemtabrutinib Final Market Formulation 2 (FMF2) in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Food on Nemtabrutinib (MK-1026) in Healthy Participants (MK-1026-017)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-017; MK-1026-17 (Other: MSD)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemtabrutinib Treatment A (Experimental): Participants receive a single dose of nemtabrutinib on Day 1 under fasted conditions (on an empty stomach after a 10-hour overnight fast)
  Interventions: Drug: Nemtabrutinib
- Nemtabrutinib Treatment B (Experimental): Participants receive a single dose of nemtabrutinib on Day 1 under fed conditions (after a high-fat meal)
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Oral Tablet
  Other Names: MK-1026; ARQ-531

SUMMARY:
The goal of the study is to learn what happens to levels of nemtabrutinib in a healthy person's body over time. Researchers will compare what happens to nemtabrutinib in the body when it is given under fasted (on an empty stomach) and fed (after a high-fat meal) conditions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

* Is in good health based on medical history, physical examination, vital signs (VS) measurements, electrocardiograms (ECGs), and laboratory safety tests performed before randomization
* Has a body mass index (BMI) 18.0 to 32.0 kg/m^2 (inclusive)

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the AUC0-inf of nemtabrutinib in plasma.

SECONDARY OUTCOMES:
Time Taken for the Drug to Appear in the Systemic Circulation Following Administration (Tlag) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Tlag of nemtabrutinib in plasma.
Apparent Terminal Elimination Half-Life (t1/2) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the t1/2 of nemtabrutinib in plasma.
Apparent Total Plasma Clearance (CL/F) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the CL/F of nemtabrutinib in plasma.
Apparent Volume of Distribution During Terminal Elimination Phase (Vz/F) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Vz/F of nemtabrutinib in plasma.
Area Under the Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the AUC0-last of nemtabrutinib in plasma.
Maximum Observed Concentration (Cmax) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Cmax of nemtabrutinib in plasma.
Time of the Maximum Observed Concentration (Tmax) of Nemtabrutinib | Predose and at designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Tmax of nemtabrutinib in plasma.
Number of Participants Who Experience an Adverse Event (AE) | Up to 30 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue the Study Intervention Due to an AE | Up to 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorp Clinical Research Unit Inc. (Site 0001), Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/